CLINICAL TRIAL: NCT03017495
Title: A Single-center, Open-label Study to Investigate the Food Effect on the Pharmacokinetics of ACT-541468 and the Effect of Single- and Multiple-dose ACT-541468 on the Pharmacokinetics of Midazolam and Its Metabolite 1-Hydroxymidazolam in Healthy Male Subjects
Brief Title: A Clinical Study to Investigate the Potential Interactions Between Food and ACT-541468 and Between ACT-541468 and Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-078-104; 2016-003490-18 (EudraCT Number)
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: food-drug interaction; drug-drug interaction; pharmacokinetics
MeSH Terms: interventions — Midazolam; daridorexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Food effect and Drug-Drug interaction (Experimental): Treatments will be given to all subjects in the same fixed sequence: Treatment A (Day 1, single dose of midazolam, fasted), Treatment B (Day 2, single dose of ACT-541468 followed by single dose of midazolam, fasted), Treatment C (Day 4, single dose ACT-541468, fed), Treatment D (multiple doses of ACT-541468 from Day 5 to Day 8 + single dose of midazolam on Day 8, fasted).
  Interventions: Drug: Midazolam; Drug: ACT-541468

INTERVENTIONS:
Drug: Midazolam — 2 mg/mL oral solution
Drug: ACT-541468 — Hard gelatin capsules for oral use at a strength of 25 mg

SUMMARY:
The main objectives of this phase 1 trial are to evaluate the effect of food on the pharmacokinetics (i.e. how long and how much a compound is present in the blood) of ACT-541468 and to evaluate whether ACT-541468 can affect the pharmacokinetics of midazolam, a CYP3A4 substrate.

DETAILED DESCRIPTION:
Food effect will be assessed by comparing the pharmacokinetic (PK) parameters of a single dose of ACT-541468 under fasted (Treatment B) and fed (Treatment C) conditions.

Potential CYP3A4 inhibiting / inducing effects of ACT-541468 will be assessed by comparing the PK parameters of midazolam alone (Treatment A) and midazolam given with a single dose of ACT-541468 (Treatment B) or with multiple doses of ACT-541468 (Treatment D).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Male subjects aged from 18 to 45 years (inclusive) at screening
* Body mass index (BMI) from 18.0 to 30.0 kg/m2 (inclusive) at screening
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests

Exclusion Criteria:

* Any contraindication to the study treatments
* History or clinical evidence of any disease or medical / surgical condition or treatment, which may put the subject at risk of participation in the study or may interfere with the absorption, distribution, metabolism or excretion of the study treatments
* History of narcolepsy or cataplexy or modified Swiss narcolepsy scale total score < 0
* Any circumstances or conditions, which, in the opinion of the investigator, may affect the subject's full participation in the study or compliance with the protocol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-541468 | PK blood samples on Day 2, Day 4 and Day 8: before administration of ACT-541468 and up to 24 hours post-dose, and on Day 6 and Day 7: before ACT-541468 administration only
  Cmax is directly determined from the plasma concentrations-time curves of ACT-541468
Time to reach Cmax (tmax) of ACT-541468 | PK blood samples on Day 2, Day 4 and Day 8: before administration of ACT-541468 and up to 24 hours post-dose, and on Day 6 and Day 7: before ACT-541468 administration only
  Tmax is directly determined from the plasma concentrations-time curves of ACT-541468
Area under the plasma concentration-time curve [AUC(0-24)] of ACT-541468 | PK blood samples on Day 2, Day 4 and Day 8: before administration of ACT-541468 and up to 24 hours post-dose, and on Day 6 and Day 7: before ACT-541468 administration only
  AUC is calculated from time zero to 24 hours post dose
Terminal half-life (t1/2) of ACT-541468 | PK blood samples on Day 2, Day 4 and Day 8: before administration of ACT-541468 and up to 24 hours post-dose, and on Day 6 and Day 7: before ACT-541468 administration only
  t1/2 is calculated from the plasma concentrations-time curves of ACT-541468
Maximum plasma concentration (Cmax) of midazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  Cmax is directly obtained from the plasma concentrations-time curves of midazolam
Time to reach Cmax (tmax) of midazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  Tmax is directly obtained from the plasma concentrations-time curves of midazolam
Area under the plasma concentration-time curve [AUC(0-24)] of midazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  AUC is calculated from time zero to 24 hours post dose
Terminal half-life (t1/2) of midazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  t1/2 is calculated from the plasma concentrations-time curves of midazolam
Maximum plasma concentration (Cmax) of 1-hydroxymidazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  Cmax is directly determined from the plasma concentrations-time curves of 1-hydroxymidazolam
Time to reach Cmax (tmax) of 1-hydroxymidazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  Tmax is directly determined from the plasma concentrations-time curves of 1-hydroxymidazolam
Area under the plasma concentration-time curve [AUC(0-24)] of 1-hydroxymidazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  AUC is calculated from time zero to 24 hours post dose
Terminal half-life (t1/2) of 1-hydroxymidazolam | PK blood samples on Day 1, Day 2, Day 8: before administration of midazolam and up to 24 hours post dose
  t1/2 is calculated from the plasma concentrations-time curves of 1-hydroxymidazolam

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events and serious adverse events | From baseline to end-of-study, i.e.,maximum 5 days after Day 8
Maximum plasma concentration (Cmax) of ACT-541468 metabolites | PK blood samples on Day 8, before administration of ACT-541468 and up to 24 hours post dose
Time to reach Cmax (tmax) of ACT-541468 metabolites | PK blood samples on Day 8, before administration of ACT-541468 and up to 24 hours post dose
Area under the plasma concentration-time curve [AUC(0-24)] of ACT-541468 metabolites | PK blood samples on Day 8, before administration of ACT-541468 and up to 24 hours post dose
Terminal half-life (t1/2) of ACT-541468 metabolites | PK blood samples on Day 8, before administration of ACT-541468 and up to 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Boof, PhD, Study Director — Actelion
Locations (1):
- Investigator Site, Kiel, Germany